CLINICAL TRIAL: NCT02051647
Title: Copeptin as a Stress Marker During a Written Examination - the CoEXAM
Brief Title: Copeptin as a Stress Marker During a Written Examination
Acronym: CoEXAM
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 325/13
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: medical students; Basel University

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Serum, Li-Heparin
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate whether copeptin levels increase upon a psychological stress (i.e. written examination) and whether copeptin levels measured immediately before the written examination predict success of the examination.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Member of 4th year in medical course at Basel University

Exclusion Criteria:

* Intake of any medication (except birth control pill)
* BMI over 30kg/m2
* Evidence of acute disease
* History of chronic illness, including chronic psychiatric disease
* Anamnestic certain or assumed pregnancy
* Regularly smoking students

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 42 healthy voluntary medical students studying in the 4th year at Basel University
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in copeptin levels upon examination stress comparing copeptin levels prior and after examination | 4 hours

SECONDARY OUTCOMES:
Correlation between copeptin levels prior to an exam and exam success | 4 hours
Correlation to cortisol as the classical stress marker | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hopsital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Urwyler SA, Schuetz P, Sailer C, Christ-Crain M. Copeptin as a stress marker prior and after a written examination--the CoEXAM study. Stress. 2015 Jan;18(1):134-7. doi: 10.3109/10253890.2014.993966. Epub 2015 Jan 8. PMID 25472823